CLINICAL TRIAL: NCT01838603
Title: Patient Experience of Interventional Pain Management. Qualitative Study
Status: Completed | Type: Observational
Sponsor: Eques Indolor AB (Other)
Responsible Party: Sponsor
Other Study IDs: SE-Dnr-2012-446-31M-3
Record Dates: First submitted 2013-04-19; First posted 2013-04-24 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2016-09

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Interventional pain management patients: Patients passed through interventional pain management program
  Interventions: Other: Qualitative interview

INTERVENTIONS:
Other: Qualitative interview — Qualitative interview to sample the patients feelings, experiences and thoughts risen by the treatments in the program

SUMMARY:
There are quite a few qualitative studies done to find out patients experience of chronic pain. There are no studies on what the patients feel and what thoughts and feelings arise in the patients that are exposed to interventional pain management. This study aims to illuminate how it is to live through an interventional pain management program.

DETAILED DESCRIPTION:
A qualitative interview is performed with patients that have passed through an interventional pain management program. The transcribed interviews are analyzed with qualitative content analysis according to Graneheim and Lundman in order to illuminate the experience, feelings and thoughts arisen among the patients.

ELIGIBILITY:
Inclusion Criteria:

Patients passed through an interventional pain management program

Exclusion Criteria:

Purposeful sampling will be applied

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic pain
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2013-04; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Experience of interventional pain management | 1 year
  Qualitative interview performed at one occasion where the patient describes the experience of the interventional pain management he/she has passed through

CONTACTS AND LOCATIONS:
Overall Officials: Johan Hambraeus, MD, Study Director
Locations (1):
- Smärtkliniken Eques Indolor, Vallentuna, Sweden

REFERENCES:
- [Derived] Hambraeus J, Hambraeus KS, Sahlen KG. Patient perspectives on interventional pain management: thematic analysis of a qualitative interview study. BMC Health Serv Res. 2020 Jul 1;20(1):604. doi: 10.1186/s12913-020-05452-7. PMID 32611397